CLINICAL TRIAL: NCT00935987
Title: A Phase I/II, Open-Label, Dose-Escalation Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Orally-Administered CYT387 in Primary Myelofibrosis or Post-Polycythemia Vera or Post-Essential Thrombocythemia Myelofibrosis.
Brief Title: Safety and Efficacy Study of CYT387 in Primary Myelofibrosis (PMF) or Post-polycythemia Vera (PV) or Post-essential Thrombocythemia (ET)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCL09101
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis
Keywords: Primary Myelofibrosis; Post-Polycythemia Vera; Post-Essential Thrombocythemia; CYT387
MeSH Terms: conditions — Primary Myelofibrosis | interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

ARMS (1):
- CYT387 (Experimental)
  Interventions: Drug: CYT387

INTERVENTIONS:
Drug: CYT387 — For the Part 1 dose-escalation portion of the study, patients will be assigned to dose levels in successive cohorts starting with a dose in the first cohort of 100 mg/day. CYT387 will be orally self-administered as a single daily dose beginning on Day 1 of the study, and thereafter at approximately the same time each day of the 28-day cycle. It is recommended that all doses be preceded by a 2-hour fast from food and beverages, and be followed by a 1-hour post-dose fast from food and beverages.
  Twenty additional patients will be assigned to a 150 mg BID (twice daily) dosing schedule. CYT387 will be orally self-administered twice-daily with doses approximately 10-12 hours apart beginning on Day 1 of the study, and thereafter at approximately the same times each day of the 28-day cycle.
  For the Part 2 dose confirmation portion of the study, patients will be assigned to either 150 mg or 300 mg QD (once daily) dose groups.
  Other Names: Momelotinib

SUMMARY:
This study seeks to (i) determine a safe and tolerated dose of CYT387 (momelotinib) given to patients with PMF, post-PV or post-ET and, (ii) assess the effectiveness of orally-administered CYT387 as a treatment for PMF, post-PV or post-ET.

DETAILED DESCRIPTION:
The myeloproliferative neoplasms (MPN), most notably polycythemia vera (PV), essential thrombocythemia (ET), and primary myelofibrosis (PMF) are a diverse but inter-related suite of clonal disorders of pluripotent hematopoietic stem cells (Tefferi et al., 2008). The MPN share a range of biological, pathological, and clinical features including the relative overproduction of one or more cells of myeloid origin, growth factor independent colony formation in vitro, marrow hypercellularity, extramedullary hematopoiesis, splenomegaly and hepatomegaly, and thrombotic and/or hemorrhagic diatheses (Tefferi et al., 2005).

This is an open-label, non-randomized, dose-escalation study, to be conducted in two phases: a single-centre dose-escalation phase with supernumerary patient addition (Part 1), to determine the safety and tolerability of CYT387, and to identify a therapeutic dose for the confirmation portion of the study; and a multiple-centre dose-confirmation phase (Part 2), which will be a cohort expansion at or below the maximum tolerated dose (MTD) of CYT387.

In Part 1 of the study, patients will be assigned to dose levels in successive cohorts starting with a dose in the first cohort of 100 mg/day, administered orally as a single daily dose (ie QD: at least 20 and no more than 28 hours apart, preferably in a fasted state at least one hour before and two hours after a meal). Dose-escalation will proceed initially with a 1.5-fold increment however, based on toxicity and efficacy information at a specific dose level, the dose escalation increment may be reduced to a 1.25-fold escalation at the discretion of the investigator. At any dose level, if one patient experiences a Grade 2 toxicity or higher, the dose-escalation may only proceed with 1.25-fold increments.

The MTD is defined as the highest dose level at which > 2 of 6 subjects develop first cycle DLT. New dose levels may begin accrual only if all subjects at the current dose level have been observed for a minimum of 28 days from the first day of treatment. The recommended Phase II dose will be the MTD unless significant clinical activity (efficacy) is seen below the MTD. With the exception of the first cohort, dose levels may be decreased from the intended dose levels for the next cohort, if Grade 2 or greater toxicities are observed.

Twenty (20) patients will be assigned to receive CYT387 at 150 mg twice daily (BID) with doses approximately 10-12 hours apart to determine the comparative safety, tolerability and preliminary activity of CYT387 administered twice-daily. Initially, a maximum of 6 (six) patients will be enrolled for safety assessment. If none of the six patients experiences a first-cycle DLT, then the remaining 14 patients may be enrolled following approval by the Data Safety Monitoring Board (DSMB).

In the multi-centre portion of the study (Part 2), sixty (60) additional patients will be dosed at either 150 mg or 300 mg once daily (QD). Subjects will be evaluated weekly for the first cycle, every 2 weeks for cycle 2, and at the end of each subsequent cycle for up to 9 cycles of CYT387 treatment. If, after 6 months of therapy an individual patient has not experienced a drug-related serious adverse event (SAE), the investigator may, with the written concurrence of the independent safety monitor, elect to have that patient's monthly safety assessment performed by a registered medical practitioner remote to the investigational centre. Subjects will return for a follow-up visit 30 days after completion of the last dose of study drug. Subjects who achieve at least stable disease or better and tolerate the drug well may be allowed to continue to receive CYT387 beyond the planned 9 cycles under the extension protocol CCL09101E.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PMF or post-polycythemia Vera (PV) or post-essential Thrombocythemia (ET) MF as per revised World Health Organization (WHO) criteria.
* High-risk or Intermediate-2 risk MF (as defined by the International Prognostic Scoring System [IPSS]; Appendix 13.6); or intermediate-I risk MF (IPSS) associated with symptomatic splenomegaly/hepatomegaly and/or unresponsive to available therapy.
* Must be at least 18 years of age with life expectancy of ≥ 12 weeks.
* Must be able to provide informed consent and be willing to sign an informed consent form.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Must have evidence of acceptable organ function within 7 days of initiating study drug as evidenced by the following:

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN) (or ≤ 5 x ULN if in the investigator's opinion the elevation is due to extramedullary hematopoiesis)
  * Bilirubin ≤ 2.0 x ULN or direct bilirubin < 1.0
  * Serum creatinine ≤ 2.5 x ULN
  * Absolute neutrophil count ≥ 500/µL
  * Platelet count ≥ 50,000/µL
* Females of childbearing potential must have a negative pregnancy test within 4 days of initiating study drug.

Exclusion Criteria:

* Any chemotherapy (eg, hydroxyurea), immunomodulatory drug therapy (eg, thalidomide), immunosuppressive therapy, corticosteroids > 10 mg/day prednisone or equivalent, or growth factor treatment (eg, erythropoietin) within 14 days prior to initiation of study drug.
* Incomplete recovery from major surgery within four weeks of study entry.
* Radiation therapy within four weeks of study entry.
* Women of childbearing potential, unless surgically sterile for at least 3 months (ie, hysterectomy), OR postmenopausal for at least 12 months (FSH > 30 U/mL), OR unless they agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through end of study. Permitted methods for preventing pregnancy must be communicated to study subjects and their understanding confirmed.
* Men who partner with a woman of childbearing potential, unless they agree to take appropriate precautions to avoid pregnancy (with at least 99% certainty) from screening through to the end of study. Permitted methods for preventing pregnancy must be communicated to study subjects and their understanding confirmed.
* Females who are pregnant or are currently breastfeeding.
* Known positive status for HIV.
* Clinically active hepatitis B or C.
* Diagnosis of another malignancy unless free of disease for at least three years following therapy with curative intent. Patients with early-stage basal cell or squamous cell skin cancer, cervical intraepithelial neoplasia, cervical carcinoma in situ or superficial bladder cancer may be eligible to participate at the Investigator's discretion.
* Any acute active infection.
* Cardiac dysrhythmias requiring treatment, or prolongation of the QTc (Fridericia) interval to > 450 msec for males or > 470 msec for females at prestudy screening, unless attributable to pre-existing bundle branch block.
* Presence of ≥ Grade 2 peripheral neuropathy.
* Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), uncontrolled or unstable angina, myocardial infarction, cerebrovascular accident, or pulmonary embolism within 3 months prior to initiation of study drug.
* Uncontrolled inter current illness or any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, dose-limiting toxicities (DLTs) and maximum tolerated dose (MTD) of orally-administered CYT387 in patients with PMF or post-ET/PV MF. | Ongoing throughout therapy up until 30 days after last dose of CYT387
Objective Response Rate (ORR), as measured by complete response (CR) rate, partial response (PR) rate and clinical improvement (CI) rate according to International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) consensus criteria | Baseline to study completion
  The Objective Response Rate (ORR), as measured by complete response (CR) rate, partial response (PR) rate and clinical improvement (CI) rate according to International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) is to be measured at the end of every cycle of therapy.
Pharmacokinetics of CYT387 in patients with PMF or post-ET/PV MF | Baseline to end of Cycle 1
  The pharmacokinetics (PK) of CYT387 in patients with PMF or post-ET/PV MF is to be assessed on Day 1 and Day 28 in Cycle 1 of therapy

SECONDARY OUTCOMES:
Effect of CYT387 on bone marrow or peripheral blood cytogenetic findings in patients with PMF or post-ET/PV MF. | Baseline to study completion
  The effect of CYT387 on bone marrow or peripheral blood cytogenetic findings in patients with PMF or post-ET/PV MF is to be assessed at the end of every third cycle of therapy.
Effect of CYT387 on peripheral blood granulocyte JAK2V617F allele burden in patients with PMF or post-ET/PV MF. | Baseline to study completion
  The effect of CYT387 on peripheral blood granulocyte JAK2V617F allele burden in patients with PMF or post-ET/PV MF is to be assessed at the end of each cycle of therapy (in relevant patients only)
Effect of CYT387 on peripheral blood endogenous myeloid colony formation in patients with PMF or post-ET/PV MF. | Baseline to study completion
  The effect of CYT387 on peripheral blood endogenous myeloid colony formation in patients with PMF or post-ET/PV MF is to be assessed at the end of each cycle of therapy.
Effect of CYT387 on plasma levels of inflammatory, fibrogenic and angiogenic cytokines in patients with PMF or post-ET/PV MF | Baseline to study completion
  The effect of CYT387 on plasma levels of inflammatory, fibrogenic and angiogenic cytokines in patients with PMF or post-ET/PV MF is to be assessed at the end of each cycle of therapy.
Pharmacodynamic correlates of CYT387 activity in patients with PMF or post-ET/PV MF who are receiving treatment with CYT387. | Baseline to Cycle 9
  The pharmacodynamic correlates of CYT387 activity in patients with PMF or post-ET/PV MF who are receiving treatment with CYT387 are to be assessed on Day 1 of Cycles 1, 3, 6 and 9.

CONTACTS AND LOCATIONS:
Overall Officials: Ayalew Tefferi, MD, Study Chair — Mayo Clinic; Andrew Roberts, MD, Principal Investigator — Melbourne Health; Jason Gotlib, MD, Principal Investigator — Stanford University; Vikas Gupta, MD, Principal Investigator — Princess Margaret Hospital, Canada; Shireen Sirhan, MD, Principal Investigator — Jewish General Hospital; Animesh Pardanani, MD, Principal Investigator — Mayo Clinic; Martha Wadleigh, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (3):
  - Stanford Cancer Center, Stanford, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
- The Royal Melbourne Hospital, Parkville, Victoria, Australia
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Tefferi A, Barraco D, Lasho TL, Shah S, Begna KH, Al-Kali A, Hogan WJ, Litzow MR, Hanson CA, Ketterling RP, Gangat N, Pardanani A. Momelotinib therapy for myelofibrosis: a 7-year follow-up. Blood Cancer J. 2018 Mar 7;8(3):29. doi: 10.1038/s41408-018-0067-6. PMID 29515114